CLINICAL TRIAL: NCT02318693
Title: A Randomized, Open-label, Comparative Clinical Trial to Study the Efficacy of Sitagliptin and Glibenclamide in a Short Term Treatment on the Daily Glucose Variability Using Continuous Glucose Monitoring (CGM) in Japanese Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Sitagliptin and Glibenclamide on the Glucose Variability in Japanese Participants With Type 2 Diabetes Mellitus (MK-0431-355)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-355; 152867 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin 50 mg (Experimental): Sitagliptin 50 mg administered orally once daily before breakfast for 14 days.
  Interventions: Drug: Sitagliptin
- Glibenclamide 2.50 mg TDD (Active Comparator): Glibenclamide 1.25 mg administered orally twice daily (2.5 mg TDD) for 14 days. TDD = Total daily dose.
  Interventions: Drug: Glibenclamide

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 50 mg orally once a day before breakfast for 14 days
  Other Names: MK-0431
  Arms: Sitagliptin 50 mg
Drug: Glibenclamide — Glibenclamide 1.25 mg orally twice a day (2.5 mg/day) before breakfast and dinner for 14 days
  Arms: Glibenclamide 2.50 mg TDD

SUMMARY:
This is a study of the efficacy of sitagliptin and glibenclamide in a short-term treatment on the glucose variability using continuous glucose monitoring (CGM) in Japanese participants with type 2 diabetes mellitus (T2DM). The primary hypothesis is that treatment with sitagliptin will be superior to treatment with glibenclamide in the change from baseline in mean amplitude of glycemic excursions (MAGE) through continuous glucose monitoring (CGM) after 13 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants with a diagnosis of Type 2 diabetes mellitus

Exclusion Criteria:

* History of Type 1 diabetes mellitus or ketoacidosis
* History of insulin or thiazolidinedione (including fixed-dose drug combinations containing one of these drugs) in the 12 weeks before study participation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2015-12-15 (Actual); Study Completion 2015-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Suzuki R, Eiki JI, Moritoyo T, Furihata K, Wakana A, Ohta Y, Tokita S, Kadowaki T. Effect of short-term treatment with sitagliptin or glibenclamide on daily glucose fluctuation in drug-naive Japanese patients with type 2 diabetes mellitus. Diabetes Obes Metab. 2018 Sep;20(9):2274-2281. doi: 10.1111/dom.13364. Epub 2018 Jun 11. PMID 29770541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening for study inclusion was performed over a 4-week period. Adults with type 2 diabetes were randomized into the study.
Period: Overall Study
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Started | 26 | 27
Treated | 26 | 26 (1 randomized participant did not receive treatment.)
Completed | 26 | 26
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data is provided for the Full Analysis Set (FAS) population consisting of all randomized participants who received at least one dose of study treatment, with at least one post-randomization/post-treatment observation for analysis, and with applicable baseline data.
Groups:
- Glibenclamide 2.50 mg TDD: Glibenclamide 1.25 mg administered orally twice daily (2.5 mg TDD) for 14 days.
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.2 (8.4) | 59.5 (10.7) | 59.8 (9.5)
Age, Customized [Number; unit: Participants]
  <65 years | 15 | 16 | 31
  >=65 years | 11 | 10 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 26 | 25 | 51
Body Weight [Mean (Standard Deviation); unit: kg] | 70.2 (8.2) | 70.7 (11.2) | 70.5 (9.7)
Height [Mean (Standard Deviation); unit: cm] | 169.5 (5.4) | 169.3 (5.3) | 169.4 (5.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 24.4 (2.1) | 24.6 (3.0) | 24.5 (2.6)
Duration of Diabetes Mellitus [Mean (Standard Deviation); unit: Years] | 6.4 (5.4) | 9.9 (5.5) | 8.2 (5.7)
Smoking Status [Number; unit: Participants]
  Current Smoker | 8 | 9 | 17
  Ex-Smoker | 10 | 10 | 20
  Never Smoked | 8 | 7 | 15
Alcohol Consumption [Number; unit: Drinks/week]
  0 | 8 | 5 | 13
  1 to 4 | 9 | 13 | 22
  >5 | 9 | 8 | 17
Hemoglobin A1C (HbA1C) [Mean (Standard Deviation); unit: %] — Glycosylated HbA1c is a surrogate marker of long-term glycemic control. The permissible range for study inclusion was ≥ 7.0% and < 9.0% (National Glycohemoglobin Standardization program; NGSP) at Week -2.
  % | 7.7 (0.5) | 7.9 (0.6) | 7.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Amplitude of Glycemic Excursions (MAGE) at Day 13
Description: MAGE is a popular metric for assessment of major (e.g., postprandial) glucose swings. MAGE is calculated as the average of differences between consecutive glucose peaks and nadirs greater than 1 standard deviation (SD) of 24-hour mean glucose. In this assessment, glucose levels were determined using continuous glucose monitoring (CGM) over 24 hours at Baseline and Day 13; CGM values were further corrected for blood glucose values obtained via participant-administered finger-stick. Least squares (LS) means values were derived from a constrained longitudinal analysis model. A negative (-) change from Baseline to Day 13 indicates improvement of the assessed outcome.
Time Frame: Baseline (Day -2) and Day 13
Population: The FAS population consisting of all randomized participants who received at least one dose of study treatment, with at least one post-randomization/post-treatment observation for the analysis, and with applicable baseline data was used for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Number analyzed (Participants) | 26 | 26
mg/dL | -18.5 [-30.0 to -7.1] | -9.7 [-21.1 to 1.6]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.245, constrained longitudinal analysis model; Model included terms for treatment, time and time-by-treatment interaction with a constraint that mean baseline is the same for both treatment groups; LS Means Difference = -8.8, 95% CI 2-sided [-23.8 to 6.2]

2. Secondary Outcome: Change From Baseline in the Standard Deviation of Blood Glucose Levels
Description: SD is a popular metric for assessment of postprandial glucose swings. The SD of all glycemic excursions over 24 hours (i.e., total of 288 glucose values over 24 hours) was determined for Baseline and Day 13. Original values were obtained using CGM and corrected for blood glucose values obtained via participant-administered finger-stick. LS mean values were derived from a constrained longitudinal analysis model. A negative (-) change from Baseline to Day 13 indicates improvement of the assessed outcome.
Time Frame: Baseline (Day -2) and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Number analyzed (Participants) | 26 | 26
mg/dL | -10.2 [-14.4 to -6.0] | -4.2 [-8.4 to -0.1]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.029, constrained longitudinal analysis model; [statistical method as in outcome 1, analysis 1]; LS Means Difference = -5.9, 95% CI 2-sided [-11.3 to -0.6]

3. Secondary Outcome: Change From Baseline in Maximum Incremental Postprandial Glucose Levels in Each Meal
Description: The peak postprandial glucose level during the 3 hours post meal minus the preprandial glucose level 1 hour before meal was determined for corrected CGM values at Baseline and Day 13 for breakfast, lunch, and dinner. Meals were standardized with respect to total calories, and protein, fat, and carbohydrate composition as well as timing of administration. CGM values were corrected using a participant-administered finger-stick test for blood glucose. LS mean values were derived from a constrained longitudinal analysis model. A negative (-) change from baseline to Day 13 indicates better control of postprandial glucose.
Time Frame: Baseline (Day -2) and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Number analyzed (Participants) | 26 | 26
mg/dL
  Breakfast | -24.8 [-34.1 to -15.6] | -12.0 [-21.1 to -2.9]
  Lunch | -13.2 [-24.0 to -2.3] | 1.2 [-9.6 to 11.9]
  Dinner | -9.0 [-20.9 to 2.9] | -14.1 [-25.9 to -2.3]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change from Baseline in Maximum Incremental Postprandial Glucose Levels at Breakfast. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.041, constrained longitudinal analysis model; [statistical method as in outcome 1, analysis 1]; LS Means Difference = -12.8, 95% CI 2-sided [-25.1 to -0.5]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change from Baseline in Maximum Incremental Postprandial Glucose Levels at Lunch. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.043, constrained longitudinal analysis model; [statistical method as in outcome 1, analysis 1]; LS Means Difference = -14.3, 95% CI 2-sided [-28.1 to -0.5]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change from Baseline in Maximum Incremental Postprandial Glucose Levels at Dinner. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.509, constrained longitudinal analysis model; [statistical method as in outcome 1, analysis 1]; LS Means Difference = 5.1, 95% CI 2-sided [-10.3 to 20.4]

4. Secondary Outcome: Change From Baseline in 24-hour Mean Glucose Level
Description: The mean glucose level over 24-hours at Baseline and Day 13 was determined using CGM values corrected for participant-administered finger-stick values. LS mean values were derived from a constrained longitudinal analysis model. A negative (-) change from Baseline to Day 13 indicates improvement of the assessed outcome.
Time Frame: Baseline (Day -2) and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Number analyzed (Participants) | 26 | 26
mg/dL | -19.1 [-28.5 to -9.7] | -34.8 [-44.0 to -25.5]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.020, constrained longitudinal analysis model; [statistical method as in outcome 1, analysis 1]; LS Means Difference = 15.7, 95% CI 2-sided [2.5 to 28.8]

5. Secondary Outcome: Change From Baseline in Percentage of Hypoglycemic Values (Glucose Sensor Readings: < 70, <60, <50 mg/dL)
Description: Hypoglycemia, defined as low blood glucose, is a common side effect of medications used to treat diabetes mellitus type 2. The percentage of hypoglycemic corrected CGM readings (sensor glucose <70, <60, <50 mg/dL) over a 24-hour period were determined at baseline and Day 13. CGM values were corrected using a participant-administered finger-stick test for blood glucose. LS mean values were derived from a constrained longitudinal analysis model. A negative (-) change from baseline to Day 13 indicates improvement in occurrence of hypoglycemia.
Time Frame: Baseline (Day -2) and Day 13
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Number analyzed (Participants) | 26 | 26
Percent change
  <70 mg/dL | -0.3 [-1.6 to 1.0] | 0.8 [-0.5 to 2.1]
  <60 mg/dL | -0.4 [-1.3 to 0.5] | 0.2 [-0.7 to 1.1]
  <50 mg/dL | -0.3 [-0.8 to 0.2] | -0.3 [-0.7 to 0.2]
Statistical Analysis 1: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change in Baseline in Percentage of Hypoglycemic Values < 70 mg/dL. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.134, constrained longitudinal analysis model; LS Means Difference = -1.1, 95% CI 2-sided [-2.5 to 0.3]
Statistical Analysis 2: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change in Baseline in Percentage of Hypoglycemic Values < 60 mg/dL. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.226, constrained longitudinal analysis model; LS Means Difference = -0.6, 95% CI 2-sided [-1.5 to 0.4]
Statistical Analysis 3: Comparison: Sitagliptin 50 mg vs Glibenclamide 2.50 mg TDD; Comparison: Change in Baseline in Percentage of Hypoglycemic Values < 50 mg/dL. The comparison was conducted at the α=0.05 (2-sided) significance level; Test type: Superiority or Other; p = 0.332, constrained longitudinal analysis model; LS Means Difference = 0.0, 95% CI 2-sided [-0.1 to 0.0]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: The All Subjects as Treated (ASaT) population consisting of all participants who received at least one dose of study treatment was used for analysis of safety.
Arm/Group | Sitagliptin 50 mg | Glibenclamide 2.50 mg TDD
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 11/26 | 10/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin 50 mg (N=26) | Glibenclamide 2.50 mg TDD (N=26)
Periodontitis (Infections and infestations) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (5) | 3 (4)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 10 (10) | 6 (6)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential may be deleted prior to submission; this confidentiality does not include efficacy and safety results.